CLINICAL TRIAL: NCT01802281
Title: A Randomized Trial of Vaginal Surgery for Uterovaginal Prolapse: Vaginal Hysterectomy With Native Tissue Vault Suspension vs. Mesh Hysteropexy Suspension
Brief Title: Study of Uterine Prolapse Procedures - Randomized Trial
Acronym: SUPeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PFDN-24P01
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Uterovaginal Prolapse

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hysteropexy (Active Comparator): Uphold® LITE
  Interventions: Procedure: Uphold® LITE
- Hysterectomy and USLS (Active Comparator): Vaginal hysterectomy and uterosacral ligament suspension (USLS)
  Interventions: Procedure: Uterosacral ligament suspension

INTERVENTIONS:
Procedure: Uterosacral ligament suspension — The USLS procedure used in this protocol is a modification of the technique described by Shull.
  Arms: Hysterectomy and USLS
Procedure: Uphold® LITE — The Uphold® procedure used in this protocol is a modification of the technique described by Vu and Goldberg.
  Arms: Hysteropexy

SUMMARY:
The primary purpose of this randomized clinical trial is to compare the effectiveness and safety of two transvaginal apical suspension strategies for uterovaginal prolapse: a mesh augmented hysteropexy versus vaginal hysterectomy and uterosacral ligament suspension (USLS). The primary aim is to determine whether treatment success in women who undergo the above strategies differ at time points through 3 years.

A supplemental study investigates anterior vaginal wall movement resulting from descent or rotation of the vaginal apex and/or anterior vaginal elongation, in women in both of the study arms of SUPeR.

DETAILED DESCRIPTION:
The study population will be adult women (>21 years of age) with symptomatic uterovaginal prolapse at or beyond the hymen who desire vaginal surgical management. This study is intended to be done only on women who have completed child-bearing and have an inactive uterus, defined as amenorrhea for 1 year. Therefore women will be postmenopausal or will have amenorrhea from an endometrial ablation. Amenorrhea caused from exogenous steroids, or hypothalamic disorders will not allow inclusion.

Participants will be obtained from the clinic population of each of the eight Pelvic Floor Disorders Network (PFDN) sites. Participants will be randomly assigned to have either vaginal hysterectomy and USLS or mesh hysteropexy suspension for treatment of their uterovaginal prolapse. The surgical assignment will be revealed in the operating room, after the participant is under anesthesia.

Participants will be followed for at least 36-months (3-years) post surgery and up to a maximum of 60-months (5-years) during the primary trial. Participants who complete the primary trial will be approached for consent for long-term follow-up as part of a study extension and will be followed up to a maximum of 120-months (10-years). Follow-up data will be obtained during in-person clinic visits, and study staff who are masked to the surgical assignment will be the primary person who obtain follow-up data. Although the primary study outcome does not depend on masked participants and blinded evaluators, several important participant reported secondary aims are subject to reporting bias if the participant is aware of her study assignment. Therefore, study participants, coordinators, and nurses will be masked to the study assignment. Study surgeons and anatomic evaluators will be unmasked. Evaluators conducting the POPQ exam will be a co-investigator, fellow or other qualified nurse who did not perform the study surgery.

Surgical failure rates will be compared using survival analysis approaches appropriate for interval censored data (classic log-rank tests and survival models using a generalized linear model approach with a complementary log-log link) and secondary outcomes will be reported as rates in each group or as group means and evaluated with the appropriate parametric or nonparametric statistical tests.

Throughout the study, the PFDN Data Safety and Monitoring Committee (DSMB) will review study data and decide if the study can or cannot continue. Additionally, this study will adhere to the CONSORT guidelines for performing and reporting randomized controlled trials (Begg et al 1996). Women who are eligible but decline enrollment will be characterized in a manner consistent with CONSORT requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 21 or older who have completed child -bearing
2. Prolapse beyond the hymen (defined as Ba, Bp, or C > 0 cm)
3. Uterine descent into at least the lower half of the vagina (defined as point C> -TVL/2) )
4. Bothersome bulge symptoms as indicated on question 3 of the PFDI-20 form relating to 'sensation of bulging' or 'something falling out'
5. Desires vaginal surgical treatment for uterovaginal prolapse
6. Available for up to 60 month follow-up
7. Amenorrhea for the past 12 months from either menopause or endometrial ablation
8. Not pregnant, not at risk for pregnancy or agree to contraception if at risk for pregnancy (only applicable to the rare endometrial ablation patient)
9. Eligible for no cervical cancer screening for at least 3 years

Exclusion Criteria:

1. Previous synthetic material (placed vaginally or abdominally) to augment POP repair
2. Known previous uterosacral or sacrospinous uterine suspension
3. Known adverse reaction to synthetic mesh or biological grafts; these complications include but are not limited to erosion, fistula, or abscess
4. Chronic pelvic pain
5. Pelvic radiation
6. Cervical elongation- defined as an expectation that the C point would be Stage 2 or greater postoperatively if a hysteropexy was performed. (Note: cervical shortening or trachelectomy is not an allowed intraoperative procedure within the hysteropexy treatment group).
7. Women at increased risk of cervical dysplasia requiring cervical cancer screening more often than every 3 years (e.g. HIV+ status, immunosuppression because of transplant related medications, Diethylstilbestrol (DES) exposure in utero, or previous treatment for cervical intraepithelial neoplasia (CIN)2, CIN3, or cancer)
8. Uterine abnormalities (symptomatic uterine fibroids, polyps, endometrial hyperplasia, endometrial cancer, or any uterine disease that precluded prolapse repair with uterine preservation in the opinion of the surgeon
9. Indication for ovarian removal (adnexal mass, BRCA 1/2 positivity, family history of ovarian cancer)
10. Current condition of amenorrhea caused by exogenous sex steroids or hypothalamic conditions.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Nager, MD, Principal Investigator — University of California at San Diego, UCSD Women's Pelvic Medicine Center; Anthony G Visco, MD, Principal Investigator — Duke University, Duke Division of Urogynecology and Reconstructive Pelvic Surgery; Heidi Harvie, MD, Principal Investigator — University of Pennsylvania; Marie Paraiso, MD, Principal Investigator — Cleveland Clinic, Department OB/GYN; Charles R Rardin, MD, Principal Investigator — Brown/ Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery; Holly E Richter, PhD, MD, Principal Investigator — University of Alabama at Birmingham, Department of Obstetrics and Gynecology; Kate Meriwether, MD, Principal Investigator — University of New Mexico Health Sciences Center, Department of Obstetrics and Gynecology; Halina M Zyczynski, MD, Principal Investigator — Magee-Women's Hospital, Department of Obstetrics and Gynecology; Sonia Thomas, DrPH, Principal Investigator — RTI International
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Department of Obstetrics and Gynecology, Birmingham, Alabama
  - University of California at San Diego, UCSD Women's Pelvic Medicine Center, La Jolla, California
  - University of New Mexico Health Sciences Center, Department of Obstetrics and Gynecology, Albuquerque, New Mexico
  - Duke University, Duke Division of Urogynecology and Reconstructive Pelvic Surgery, Durham, North Carolina
  - Cleveland Clinic, Department OB/GYN, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee-Women's Hospital, Department of Obstetrics and Gynecology, Pittsburgh, Pennsylvania
  - Brown/ Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bradley MS, Sridhar A, Ferrante K, Andy UU, Visco AG, Florian-Rodriguez ME, Myers D, Varner E, Mazloomdoost D, Gantz MG; NICHD Pelvic Floor Disorders Network. Association Between Enlarged Genital Hiatus and Composite Surgical Failure After Vaginal Hysterectomy With Uterosacral Ligament Suspension. Urogynecology (Phila). 2023 May 1;29(5):479-488. doi: 10.1097/SPV.0000000000001309. Epub 2022 Dec 23. PMID 36701331
- [Derived] Napoe GS, Luchristt D, Sridhar A, Ellington D, Ridgeway B, Mazloomdoost D, Sung V, Ninivaggio C, Harvie H, Santiago-Lastra Y, Gantz MG, Zyczynski HM. Reoperation for prolapse recurrence after sacrospinous mesh hysteropexy: characteristics of women choosing retreatment. Int Urogynecol J. 2023 Jan;34(1):255-261. doi: 10.1007/s00192-022-05411-2. Epub 2022 Nov 30. PMID 36449027
- [Derived] Nager CW, Visco AG, Richter HE, Rardin CR, Komesu Y, Harvie HS, Zyczynski HM, Paraiso MFR, Mazloomdoost D, Sridhar A, Thomas S; National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Effect of sacrospinous hysteropexy with graft vs vaginal hysterectomy with uterosacral ligament suspension on treatment failure in women with uterovaginal prolapse: 5-year results of a randomized clinical trial. Am J Obstet Gynecol. 2021 Aug;225(2):153.e1-153.e31. doi: 10.1016/j.ajog.2021.03.012. Epub 2021 Mar 12. PMID 33716071
- [Derived] Lukacz ES, Sridhar A, Chermansky CJ, Rahn DD, Harvie HS, Gantz MG, Varner RE, Korbly NB, Mazloomdoost D; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network (PFDN). Sexual Activity and Dyspareunia 1 Year After Surgical Repair of Pelvic Organ Prolapse. Obstet Gynecol. 2020 Sep;136(3):492-500. doi: 10.1097/AOG.0000000000003992. PMID 32769645
- [Derived] Nager CW, Visco AG, Richter HE, Rardin CR, Rogers RG, Harvie HS, Zyczynski HM, Paraiso MFR, Mazloomdoost D, Grey S, Sridhar A, Wallace D; NICHD Pelvic Floor Disorders Network. Effect of Vaginal Mesh Hysteropexy vs Vaginal Hysterectomy With Uterosacral Ligament Suspension on Treatment Failure in Women With Uterovaginal Prolapse: A Randomized Clinical Trial. JAMA. 2019 Sep 17;322(11):1054-1065. doi: 10.1001/jama.2019.12812. PMID 31529008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hysteropexy | Hysterectomy and USLS
Started (Started indicates randomized into the SUPeR study) | 93 | 90
Eligible and Received Randomized Treatment (A small number of randomized participants received the randomized treatment but were found to be ineligible for the intervention) | 88 | 87
Completed Year 1 Follow-up | 88 | 86
Completed Year 2 Follow-up | 87 | 84
Completed (Completed Year 3 Follow-up) | 85 | 84
Not Completed | 8 | 6
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Ineligible | 5 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all randomized participants that received the assigned intervention and were determined to still be eligible for the intervention after review of the initial POP-Q and PFDI-20.
Groups:
- UPHOLD: UPHOLD Procedure
- USLS: Vaginal hysterectomy and Uterosacral Ligament Suspension (USLS)
- Total: Total of all reporting groups
Arm/Group | UPHOLD | USLS | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (7) | 66.2 (7) | 65.9 (7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 88 | 87 | 175
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 0 | 4 | 4
  Asian | 2 | 1 | 3
  Black/African American | 8 | 3 | 11
  More than one race | 0 | 1 | 1
  Other | 5 | 1 | 6
  White | 73 | 77 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latina | 9 | 7 | 16
  Not Hispanic/Not Latina | 76 | 78 | 154
  Unknown/Not Reported | 3 | 2 | 5
Marital Status [Count of Participants; unit: Participants]
  Divorced, separated | 16 | 13 | 29
  Married/Living with partner | 56 | 58 | 114
  Single | 9 | 7 | 16
  Widowed | 7 | 9 | 16
Education [Count of Participants; unit: Participants]
  4-year College Degree | 16 | 20 | 36
  Associate College Degree | 22 | 19 | 41
  Graduate Degree | 11 | 15 | 26
  High School/GED | 31 | 26 | 57
  Less than High School | 6 | 5 | 11
  Unknown/Not Reported | 2 | 2 | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (4.0) | 28.2 (4.4) | 28.5 (4.2)
Current Smoker [Count of Participants; unit: Participants]
  No | 85 | 86 | 171
  Yes | 3 | 1 | 4
Number of Pregnancies [Median (Full Range); unit: Number of pregnancies] | 3 [0 to 12] | 3 [0 to 7] | 3 [0 to 12]
Number of Vaginal Deliveries [Median (Full Range); unit: Number of deliveries] | 3 [0 to 10] | 2 [0 to 6] | 3 [0 to 10]
Menstrual Status [Count of Participants; unit: Participants]
  pre-menopausal (includes peri-menopausal)/not sure | 2 | 2 | 4
  post-menopausal (no menses for the last 12-months) | 86 | 85 | 171
POP-Q Ba [Mean (Standard Deviation); unit: cm] — Pelvic Organ Prolapse Quantification System (POP-Q) Point Ba represents the most distal (i.e. most dependent) position of any part of the upper anterior vaginal wall (between the vaginal cuff or anterior vaginal fornix and Point Aa). Point Ba coincides with Point Aa (-3 cm) in a woman who has no anterior POP. In a woman with severe POP, Ba coincides with Point C.
  cm | 3.3 (2.0) | 3 (2.2) | 3.1 (2.1)
POP-Q Bp [Mean (Standard Deviation); unit: cm] — POP-Q Point Bp represents the most distal position of any part of the upper posterior vaginal wall (between the vaginal cuff or posterior vaginal fornix and Point Ap).
  cm | 0.4 (3.0) | 0.7 (3.0) | 0.6 (3.0)
POP-Q C [Mean (Standard Deviation); unit: cm] — POP-Q Point C is measured in cm relative to the hymen with negative values being proximal to the hymen and positive values distal to the hymen. Point C represents either the most distal edge of the cervix or the leading edge of the vaginal cuff after total hysterectomy.
  cm | 0.4 (3.5) | 0.7 (3.6) | 0.5 (3.5)
POP-Q TVL [Mean (Standard Deviation); unit: cm] — The POP-Q TVL (total vaginal length) is the length of the vagina (cm) from posterior fornix to hymen when Point C or D is reduced to its full normal position.
  cm | 9.1 (1.1) | 9.1 (1.1) | 9.1 (1.1)
POP-Q Stage [Count of Participants; unit: Participants] — The POP-Q is summarized by stages in which higher stages indicate worse prolapse:
  Stage 0: No prolapse is demonstrated.
  Stage 1: The most distal portion of the prolapse is more than 1 cm above the level of the hymen.
  Stage 2: The most distal portion of the prolapse is between 1 cm above the hymen and 1 cm below the hymen.
  Stage 3: The most distal portion of the prolapse is more than 1 cm beyond the plane of the hymen, but not further than 2 cm less than the TVL.
  Stage 4: Complete eversion or eversion to within 2 cm of the TVL.
  Participants
    2 | 15 | 19 | 34
    3 | 63 | 59 | 122
    4 | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Failure
Description: Failure was defined as any of the following: retreatment for prolapse, any POP-Q measure beyond the hymen, or presence of bother on PFDI vaginal bulge question. Under the permanent failure state assumption, the number of participants shown at each visit includes all participants who were still participating in the study or had a failure outcome prior their withdrawal. Similarly, the denominator number of participants for the cumulative failure at each visit includes all participants who were still participating in the study and attended the visit or had any failure outcome prior their withdrawal or missed visit.
Time Frame: 6 Months through 36 Months
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and received the assigned treatment. Participants were included at each time point at which they provided outcome data after baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
Participants
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months: Non-Failure | 78 | 69
  6 Months: Failure | 9 | 16
  12 Months: number analyzed (Participants) | 86 | 85
  12 Months: Non-Failure | 71 | 63
  12 Months: Failure | 15 | 22
  18 Months: number analyzed (Participants) | 85 | 84
  18 Months: Non-Failure | 66 | 58
  18 Months: Failure | 19 | 26
  24 Months: number analyzed (Participants) | 80 | 83
  24 Months: Non-Failure | 59 | 54
  24 Months: Failure | 21 | 29
  30 Months: number analyzed (Participants) | 79 | 83
  30 Months: Non-Failure | 55 | 52
  30 Months: Failure | 24 | 31
  36 Months: number analyzed (Participants) | 79 | 81
  36 Months: Non-Failure | 53 | 47
  36 Months: Failure | 26 | 34

2. Secondary Outcome: At-visit Failure
Description: Failure was defines as any of the following: retreatment for prolapse, any POP-Q measure beyond the hymen, or presence of bother on PFDI vaginal bulge question. Under the transient failure state assumption, the number of participants shown at each visit includes all participants who were still participating in the study. Similarly, the denominator number of participants for the transient failure at each visit includes all participants who were still participating in the study and attended the visit or who missed the visit but had a retreatment failure outcome prior to their missed visit.
Time Frame: 6 months through 36 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
Participants
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months: Non-failure | 78 | 69
  6 Months: Failure | 9 | 16
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months: Non-failure | 74 | 65
  12 Months: Failure | 12 | 19
  18 Months: number analyzed (Participants) | 84 | 83
  18 Months: Non-failure | 69 | 65
  18 Months: Failure | 15 | 18
  24 Months: number analyzed (Participants) | 79 | 80
  24 Months: Non-failure | 64 | 63
  24 Months: Failure | 15 | 17
  30 Months: number analyzed (Participants) | 78 | 78
  30 Months: Non-failure | 60 | 60
  30 Months: Failure | 18 | 18
  36 Months: number analyzed (Participants) | 78 | 78
  36 Months: Non-failure | 62 | 57
  36 Months: Failure | 16 | 21

3. Other Pre Specified Outcome: Change From Baseline PFDI Score
Description: The Pelvic Floor Distress Inventory is a 20-question, validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of an overall scale (range: 0-300) comprised of 3 sub-scales: 1. Pelvic Organ Prolapse Distress Inventory (range: 0-100), 2. Colorectal Anal Distress Inventory (range: 0-100), and 3. Urinary Distress Inventory (range: 0-100). The range of responses on the CRADI is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Scores are calculated by multiplying the mean value of all questions answered by 25 for the scale. The range of responses is: 0-100 with 0 (least distress) to 100 (most distress). Lower scores indicate better function / fewer symptoms. Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -81.7 [-93.3 to -70.1] | -73 [-84.8 to -61.1]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -81.2 [-92.9 to -69.6] | -75.4 [-87.3 to -63.5]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -78.7 [-90.5 to -67] | -75.8 [-87.8 to -63.9]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -82.1 [-93.9 to -70.2] | -76.6 [-88.7 to -64.5]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -79.8 [-91.7 to -67.8] | -80.1 [-92.3 to -67.8]

4. Other Pre Specified Outcome: Change From Baseline CRADI Score
Description: as for outcome 3
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -11.5 [-15.6 to -7.4] | -11.1 [-15.3 to -6.9]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -11.1 [-15.2 to -7] | -11.2 [-15.4 to -7]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -10.6 [-14.8 to -6.5] | -11.9 [-16.1 to -7.6]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -12.4 [-16.6 to -8.2] | -11.4 [-15.7 to -7.2]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -11.4 [-15.6 to -7.2] | -11.6 [-15.9 to -7.2]

5. Other Pre Specified Outcome: Change From Baseline POPDI Score
Description: as for outcome 3
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -40.7 [-45.7 to -35.7] | -37 [-42.1 to -31.9]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -41.1 [-46 to -36.1] | -37.4 [-42.5 to -32.3]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -40.3 [-45.3 to -35.3] | -37.4 [-42.5 to -32.3]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -41.2 [-46.3 to -36.2] | -38 [-43.1 to -32.8]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -40.1 [-45.2 to -35] | -40.2 [-45.5 to -35]

6. Other Pre Specified Outcome: Change From Baseline UDI Score
Description: as for outcome 3
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -29.5 [-35.2 to -23.8] | -24.8 [-30.7 to -19]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -29.1 [-34.8 to -23.3] | -26.8 [-32.7 to -20.9]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -27.8 [-33.6 to -22] | -26.6 [-32.5 to -20.7]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -28.4 [-34.3 to -22.6] | -27.3 [-33.3 to -21.3]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -28.3 [-34.2 to -22.4] | -28.2 [-34.3 to -22.2]

7. Other Pre Specified Outcome: Change From Baseline PFIQ Score
Description: The Pelvic Floor Impact Questionnaire short form (PFIQ-7) measuring the impact of bladder, bowel, and vaginal symptoms on a woman''s daily activities, relationships and emotions is composed of 3 scales of 7 questions each: the Urinary Impact Questionnaire (UIQ; range 0-100), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; range 0-100), and the Colorectal-Anal Impact Questionnaire (CRAIQ; range 0-100). The range of responses on the CRAIQ is 0-3 with (0) Not at all, (1) Somewhat, (2) Moderately, and (3), Quite a bit. Scores are calculated by multiplying the mean value of all answered questions for a scale by 100 divided by 3. The range of responses is: 0-100 with 0 (least negative impact) to 100 (most negative impact). Lower scores indicate better function / fewer symptoms. Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -42.9 [-53.9 to -31.9] | -46.7 [-57.9 to -35.5]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -38.3 [-49.3 to -27.3] | -47.4 [-58.7 to -36.2]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -40.1 [-51.2 to -29.1] | -50.1 [-61.4 to -38.8]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -44 [-55.1 to -32.8] | -48.8 [-60.2 to -37.4]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -43.4 [-54.6 to -32.2] | -50.4 [-61.9 to -38.8]

8. Other Pre Specified Outcome: Change From Baseline CRAIQ Score
Description: as for outcome 7
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 86 | 84
  6 Months | -6.7 [-10.8 to -2.6] | -10.1 [-14.3 to -5.9]
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | -4.7 [-8.8 to -0.6] | -9.5 [-13.7 to -5.3]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -4.6 [-8.7 to -0.5] | -9.6 [-13.8 to -5.4]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -7.3 [-11.4 to -3.1] | -9.7 [-13.9 to -5.4]
  36 Months: number analyzed (Participants) | 78 | 74
  36 Months | -6.1 [-10.3 to -1.9] | -9.8 [-14.1 to -5.5]

9. Other Pre Specified Outcome: Change From Baseline POPIQ Score
Description: as for outcome 7
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 86 | 84
  6 Months | -15.7 [-20.6 to -10.9] | -18.9 [-23.9 to -13.9]
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | -14.6 [-19.4 to -9.7] | -19.5 [-24.5 to -14.5]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -15.9 [-20.8 to -11.1] | -20.1 [-25.1 to -15.1]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -15.9 [-20.8 to -11] | -19.1 [-24.1 to -14]
  36 Months: number analyzed (Participants) | 78 | 74
  36 Months | -16 [-21 to -11.1] | -19.9 [-25 to -14.8]

10. Other Pre Specified Outcome: Change From Baseline UIQ Score
Description: as for outcome 7
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -20.5 [-25.5 to -15.5] | -17.7 [-22.8 to -12.6]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -19 [-24 to -14.1] | -18.4 [-23.5 to -13.4]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -19.5 [-24.5 to -14.6] | -20.4 [-25.5 to -15.3]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -20.8 [-25.8 to -15.7] | -20.1 [-25.3 to -15]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -21.3 [-26.3 to -16.2] | -20.6 [-25.8 to -15.4]

11. Other Pre Specified Outcome: Change From Baseline Incontinence Severity Index
Description: Incontinence Severity Index measuring the severity of urinary incontinence is composed of 2 questions: frequency of leakage (0=Never,...,4=Every day/night) and amount of urine leakage (1=Drops, 2=small splashes, 3= More). The index score is calculated categorizing the product of the two responses. The range of responses is: 0 (no incontinence) to 12 (severe incontinence). Lower index scores indicate better function / fewer symptoms. Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 86 | 84
  6 Months | -2.4 [-3.2 to -1.6] | -1.3 [-2.1 to -0.6]
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | -2.1 [-2.9 to -1.3] | -1.4 [-2.2 to -0.6]
  18 Months: number analyzed (Participants) | 82 | 82
  18 Months | -2.1 [-2.9 to -1.3] | -1.3 [-2.1 to -0.5]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -1.9 [-2.7 to -1.2] | -1.4 [-2.2 to -0.6]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -1.9 [-2.7 to -1.1] | -1.6 [-2.5 to -0.8]

12. Other Pre Specified Outcome: Change From Baseline Functional Activity Scale
Description: Functional Activity Scale measuring the impact of incontinence symptoms on a woman''s daily activities is composed of 13 questions about normal and physically strenuous daily activities. The range of responses on the individual questions is (1) No difficulty,... (5) Not able to do it. Scores are calculated by subtracting from the maximum sum (5*13=65) the product of the mean response and number of questions, then dividing by the total range of sums (65 - 13 = 52) and multiplying by 100. The range of responses is: 0-100 with 0 (worse functionality) to 100 (Better functionality). Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | 6.3 [3.5 to 9] | 7.7 [4.9 to 10.5]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | 6.3 [3.6 to 9.1] | 6 [3.2 to 8.8]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | 5.8 [3 to 8.5] | 6.6 [3.8 to 9.5]
  24 Months: number analyzed (Participants) | 79 | 78
  24 Months | 4.9 [2.1 to 7.7] | 6.2 [3.3 to 9]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | 5.6 [2.8 to 8.5] | 4.8 [1.9 to 7.7]

13. Other Pre Specified Outcome: Change From Baseline Body Part Pain Scale
Description: The Body Part Pain Scale measuring the the pain experienced in the lower abdomen and pelvic region of the body is composed of 7 questions, each with a yes (1) or no (0) questions about experiencing pain followed by an intensity rating: 0 (No pain),..., 10 (Most intense). The score is calculated as the average of the responses. The range of responses is: 0-10 with 0 (No pain) to 10 (most intense pain). Lower scores indicate better function / fewer symptoms. Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6, 12, 18, 24, 30, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -0.4 [-0.6 to -0.2] | -0.3 [-0.5 to -0.1]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -0.5 [-0.7 to -0.3] | -0.3 [-0.5 to -0.1]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -0.5 [-0.7 to -0.3] | -0.3 [-0.5 to -0.1]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -0.6 [-0.8 to -0.3] | -0.3 [-0.6 to -0.1]
  30 Months: number analyzed (Participants) | 75 | 75
  30 Months | -0.5 [-0.7 to -0.3] | -0.3 [-0.5 to -0.1]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -0.5 [-0.7 to -0.3] | -0.3 [-0.5 to -0.1]

14. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Rest Score
Description: The Surgical Pain Scale measuring the post-surgical pain experienced by a subject is composed of 4 questions: Pain at Rest (range 0-10), Pain with Normal Activities (range 0-10), Pain with Exercise (range 0-10), and Intensity of Worst Pain (range 0-10). Lower scores indicate better less pain. Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -0.7 [-1.1 to -0.3] | -0.8 [-1.2 to -0.3]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -0.6 [-1 to -0.2] | -0.7 [-1.1 to -0.2]
  18 Months: number analyzed (Participants) | 83 | 82
  18 Months | -0.6 [-1 to -0.2] | -0.8 [-1.2 to -0.4]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -0.7 [-1.2 to -0.3] | -0.5 [-0.9 to -0.1]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -0.5 [-1 to -0.1] | -0.6 [-1.1 to -0.2]

15. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Normal Score
Description: as for outcome 14
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -0.9 [-1.3 to -0.4] | -0.8 [-1.3 to -0.4]
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months | -0.9 [-1.3 to -0.4] | -0.8 [-1.3 to -0.4]
  18 Months: number analyzed (Participants) | 83 | 83
  18 Months | -1 [-1.4 to -0.5] | -0.8 [-1.3 to -0.4]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -1 [-1.4 to -0.5] | -0.6 [-1 to -0.1]
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months | -0.7 [-1.2 to -0.2] | -0.7 [-1.2 to -0.2]

16. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Exercise Score
Description: as for outcome 14
Time Frame: 6, 12, 18, 24, and 36 Months
Population: AAn intent-to-treat (ITT) analysis which included all eligible participants who were randomized and received the assigned treatment. Participants were included at each time point at which they provided outcome data after baseline. This outcome measure is only calculated for individuals who reported exercising.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 53 | 52
units on a scale
  6 Months: number analyzed (Participants) | 42 | 37
  6 Months | -1 [-1.7 to -0.3] | -1.4 [-2.1 to -0.6]
  12 Months: number analyzed (Participants) | 38 | 40
  12 Months | -0.9 [-1.6 to -0.2] | -1.1 [-1.8 to -0.4]
  18 Months: number analyzed (Participants) | 36 | 35
  18 Months | -0.9 [-1.6 to -0.2] | -1.2 [-1.9 to -0.5]
  24 Months: number analyzed (Participants) | 35 | 31
  24 Months | -1 [-1.7 to -0.3] | -0.9 [-1.7 to -0.1]
  36 Months: number analyzed (Participants) | 31 | 29
  36 Months | -1.2 [-2 to -0.5] | -0.9 [-1.7 to -0.1]

17. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Worst Score
Description: as for outcome 14
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 85 | 82
  6 Months | -0.8 [-1.3 to -0.3] | -0.9 [-1.4 to -0.4]
  12 Months: number analyzed (Participants) | 85 | 83
  12 Months | -1 [-1.5 to -0.5] | -0.7 [-1.3 to -0.2]
  18 Months: number analyzed (Participants) | 82 | 82
  18 Months | -0.9 [-1.5 to -0.4] | -0.9 [-1.5 to -0.4]
  24 Months: number analyzed (Participants) | 78 | 78
  24 Months | -1 [-1.6 to -0.5] | -0.6 [-1.2 to 0]
  36 Months: number analyzed (Participants) | 75 | 74
  36 Months | -0.8 [-1.4 to -0.3] | -0.5 [-1.1 to 0]

18. Other Pre Specified Outcome: Change From Baseline Body Image Scale
Description: The Body Image Scale measuring how the subjects feel about their appearance and about any changes that may have resulted from their condition consists of 8 questions. The questions are scored from 0=Not at all,..., 3=Very much. The score is calculated by summing the responses and ranges from 0 to 24. Higher scores correspond to worse body image. Change = Month [6, 12, 18, 24, and 36] Score - Baseline Score.
Time Frame: 6, 12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
units on a scale
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months | -5 [-6.1 to -3.8] | -3.7 [-4.9 to -2.6]
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | -4.9 [-6.1 to -3.7] | -3.9 [-5.1 to -2.7]
  18 Months: number analyzed (Participants) | 83 | 82
  18 Months | -4.8 [-6 to -3.6] | -3.9 [-5.1 to -2.7]
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months | -4.8 [-6 to -3.6] | -3.8 [-5 to -2.6]
  36 Months: number analyzed (Participants) | 77 | 75
  36 Months | -4.9 [-6.1 to -3.7] | -3.8 [-5 to -2.6]

19. Other Pre Specified Outcome: Change From Baseline PISQ-IR Sexually Active Average Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. The PISQ-IR Sexually Active-Average Score (SA-AVG) ranges from 0 to 5 with higher scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 6, 12, 18, 24, and 36 months and the score at baseline.
Time Frame: 6, 12, 18, 24, and 36 Months
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and received the assigned treatment. Participants were included at each time point at which they provided outcome data after baseline. This outcome measure is only calculated for individuals who report being sexually active.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 30 | 40
units on a scale
  6 Months: number analyzed (Participants) | 26 | 30
  6 Months | 0.2 [0.1 to 0.4] | 0.3 [0.1 to 0.5]
  12 Months: number analyzed (Participants) | 26 | 29
  12 Months | 0.2 [0 to 0.4] | 0.3 [0.1 to 0.5]
  18 Months: number analyzed (Participants) | 25 | 27
  18 Months | 0.3 [0.1 to 0.4] | 0.2 [0.1 to 0.4]
  24 Months: number analyzed (Participants) | 24 | 26
  24 Months | 0.3 [0.1 to 0.5] | 0.3 [0.2 to 0.5]
  36 Months: number analyzed (Participants) | 23 | 27
  36 Months | 0.3 [0.1 to 0.5] | 0.3 [0.1 to 0.5]

20. Other Pre Specified Outcome: POP-Q Ba Measurement
Description: The Pelvic Organ Prolapse Quantification (POPQ) Point Ba represents the most distal (i.e. most dependent) position of any part of the upper anterior vaginal wall (between the vaginal cuff or anterior vaginal fornix and Point Aa). Point Ba coincides with Point Aa (-3 cm) in a woman who has no anterior POP. In a woman with severe POP, Ba coincides with Point C.
Time Frame: 12, 24, and 36 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
cm
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | -1.3 [-1.6 to -1] | -0.8 [-1.1 to -0.5]
  24 Months: number analyzed (Participants) | 78 | 80
  24 Months | -1.5 [-1.8 to -1.2] | -1.1 [-1.4 to -0.7]
  36 Months: number analyzed (Participants) | 78 | 74
  36 Months | -1.2 [-1.5 to -0.8] | -0.7 [-1 to -0.3]

21. Other Pre Specified Outcome: POP-Q Bp Measurement
Description: The Pelvic Organ Prolapse Quantification (POPQ) Point Bp represents the most distal position of any part of the upper posterior vaginal wall (between the vaginal cuff or posterior vaginal fornix and Point Ap).
Time Frame: 12, 24, and 36 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
cm
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | -1.9 [-2.2 to -1.6] | -2 [-2.2 to -1.7]
  24 Months: number analyzed (Participants) | 78 | 80
  24 Months | -1.8 [-2.1 to -1.5] | -2 [-2.2 to -1.8]
  36 Months: number analyzed (Participants) | 78 | 74
  36 Months | -1.7 [-2.1 to -1.4] | -1.8 [-2.1 to -1.5]

22. Other Pre Specified Outcome: POP-Q C Measurement
Description: The Pelvic Organ Prolapse Quantification (POPQ) Point C is measured in cm relative to the hymen with negative values being proximal to the hymen and positive values distal to the hymen. Point C represents either the most distal edge of the cervix or the leading edge of the vaginal cuff after total hysterectomy.
Time Frame: 12, 24, and 36 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
cm
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | -5.6 [-6.2 to -5] | -6.1 [-6.6 to -5.6]
  24 Months: number analyzed (Participants) | 78 | 80
  24 Months | -6 [-6.4 to -5.5] | -6.1 [-6.4 to -5.7]
  36 Months: number analyzed (Participants) | 78 | 74
  36 Months | -5.7 [-6.2 to -5.1] | -5.8 [-6.2 to -5.3]

23. Other Pre Specified Outcome: POP-Q TVL Measurement
Description: The Pelvic Organ Prolapse Quantification (POPQ) Total Vaginal Length (TVL) is the length of the vagina from posterior fornix tothe hymen when Point C or D is reduced to its full normal position.
Time Frame: 12, 24, and 36 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
cm
  12 Months: number analyzed (Participants) | 85 | 84
  12 Months | 8.5 [8.3 to 8.7] | 8 [7.7 to 8.2]
  24 Months: number analyzed (Participants) | 78 | 80
  24 Months | 8.6 [8.4 to 8.9] | 7.8 [7.5 to 8]
  36 Months: number analyzed (Participants) | 78 | 74
  36 Months | 8.5 [8.2 to 8.7] | 7.7 [7.4 to 8]

24. Other Pre Specified Outcome: PGI-I
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had improvement as indicated by a rating of 1 (very much better), 2 (much better).
Time Frame: 6,12, 18, 24, and 36 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | UPHOLD | USLS
Number analyzed (Participants) | 88 | 87
Participants
  6 Months: number analyzed (Participants) | 87 | 85
  6 Months: No improvement | 79 | 81
  6 Months: Improved | 8 | 4
  12 Months: number analyzed (Participants) | 86 | 84
  12 Months: No improvement | 75 | 76
  12 Months: Improved | 11 | 8
  18 Months: number analyzed (Participants) | 82 | 83
  18 Months: No improvement | 70 | 76
  18 Months: Improved | 12 | 7
  24 Months: number analyzed (Participants) | 79 | 79
  24 Months: No improvement | 69 | 71
  24 Months: Improved | 10 | 8
  36 Months: number analyzed (Participants) | 78 | 75
  36 Months: No improvement | 70 | 67
  36 Months: Improved | 8 | 8

ADVERSE EVENTS:
Time Frame: 36 Months
Groups:
- Hysterectomy: Vaginal hysterectomy and Uterosacral Ligament Suspension (USLS)
- Hysteropexy: UPHOLD Procedure
Arm/Group | Hysterectomy | Hysteropexy
All-Cause Mortality (participants affected / at risk) | 2/90 | 1/93
Serious Adverse Events (participants affected / at risk) | 10/90 | 10/93
Other Adverse Events (participants affected / at risk) | 73/90 | 73/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hysterectomy (N=90) | Hysteropexy (N=93)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (3)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hysterectomy (N=90) | Hysteropexy (N=93)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 13 (14) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 4 (5) | 10 (11)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Levator syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 39 (69) | 34 (59)
Vaginal infection (Infections and infestations) | 5 (5) | 3 (3)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femoral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hysteropexy mesh exposure (Injury, poisoning and procedural complications) | 0 (0) | 7 (12)
Midurethral sling mesh exposure (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Retained fragment of surgical packing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture exposure after 12 wks. (Injury, poisoning and procedural complications) | 17 (17) | 3 (3)
Ureteric kink (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
Vaginal laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 11 (11) | 19 (22)
Urethral caruncle (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 13 (13) | 19 (21)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 7 (8) | 6 (10)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 7 (8)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 2 (2) | 7 (7)
Fallopian tube prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 7 (8) | 3 (3)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Postmenopausal bleeding secondary to atrophy (Reproductive system and breast disorders) | 1 (1) | 4 (5)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal erosion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal scarring (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Vaginotomy (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vulvovaginal adhesion (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Excessive granulation tissue after 12 wks. (Skin and subcutaneous tissue disorders) | 10 (10) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT01802281/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT01802281/SAP_001.pdf
  • Informed Consent Form (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT01802281/ICF_002.pdf